CLINICAL TRIAL: NCT04499430
Title: Comparison of the Results of Premature Babies Started Complementary Feeding in Adjusted or Chronologically in Their Sixth Month
Brief Title: Comparison of the Results of Premature Babies Started Complementary Feeding
Acronym: COTROPBSCF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, H. Tolga Çelik, associate professor, Hacettepe University
Other Study IDs: KA-20053
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Premature Birth; Feeding Behavior
Keywords: complementary feeding; prematurity
MeSH Terms: conditions — Premature Birth; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Group 1: 29 weeks and six days of gestation and earlier
  Group 1a: complementary feeding began chronologically in the sixth month
  Group 1b: Complementary feeding corrected at sixth month
- 2: Group 2: Those whose gestational age is between 30 weeks and 33 weeks and sixth days
  Group 2a: complementary feeding began chronologically in the sixth month
  Group 2b: complementary feeding started in the sixth month, corrected
- 3: Group 3: Those whose gestational age is between 34 weeks and 37 weeks and sixth day
  Group 3a: complementary feeding began chronologically in the sixth month
  Group 3b: complementary feeding started in the sixth month, corrected

SUMMARY:
Neurological-developmental evaluations and developmental outcomes-diagnoses of premature babies are evaluated according to corrected postnatal age. Based on the limited evidence available, it can be concluded that complementary feeding may be an appropriate age for most premature babies who have reached at least the third month, generally corrected. However, for premature babies born at different gestational weeks, these periods have a relatively different meaning. A more accurate timeframe can be found in terms of complementary nutrition by evaluating chronological age and motor development together. More prospective observational studies are needed in this regard in premature babies. In the literature, there are not enough studies on the transition time to the most appropriate complementary diet for premature babies. The investigators planned to do this prospective observational study. In this study, patient groups will be randomly selected after appropriate matching. Premature babies participating in the study will be handled in three main groups (six subgroups in total). The data will be added to the case report forms. In addition to routine follow-ups, families will be called on the phone monthly, information about their babies' nutrition will be asked, whether there is a problem, questions of families will be answered, and information about complementary nutrition will be provided. At the end of the study, all data will be collected and entered into the SPSS database, which will be created.

DETAILED DESCRIPTION:
The transition to complementary feeding in premature babies (37 weeks and over) is recommended by both the World Health Organization (WHO) and the European Gastroenterology, Hepatology and Nutrition Association (ESPHGAN) for 4-6 months. However, a full consensus on the transition time to complementary feeding has not been achieved for premature babies. It is controversial whether premature babies (born 37th week of gestation) are corrected for complementary feeding in the sixth month or chronological sixth month. According to the known, there are no clinical studies investigating this topic in the literature.

Neurological-developmental evaluations and developmental outcomes-diagnoses of premature babies are evaluated according to corrected postnatal age. Based on the limited evidence available, it can be concluded that complementary feeding may be an appropriate age for most premature babies who have reached at least the third month, generally corrected. However, for premature babies born at different gestational weeks, these periods have a relatively different meaning. A more accurate timeframe can be found in terms of complementary nutrition by evaluating chronological age and motor development together. More prospective observational studies are needed in this regard in premature babies. In the literature, there are not enough studies on the transition time to the most appropriate complementary diet for premature babies. The investigators planned to do this prospective observational study.

In this study, patient groups will be randomly selected after appropriate matching. Premature babies participating in the study will be handled in three main groups (six subgroups in total).

Before the transition to complementary nutrition of the groups included in the study, breast milk and / or formula food, nutritional supplement (such as breast milk enhancer, protein supplement) intake will be recorded. The same polyvitamin preparation will be used for all premature babies. In accordance with the recommendation of the World Health Organization, 2 mg / kg / day standard oral iron prophylaxis will be started to all premature babies starting from the second chronological month. Immunization will be done in accordance with the national vaccination program.

The data will be added to the case report forms. In addition to routine follow-ups, families will be called on the phone monthly, information about their babies' nutrition will be asked, whether there is a problem, questions of families will be answered, and information about complementary nutrition will be provided. At the end of the study, all data will be collected and entered into the SPSS database, which will be created.

ELIGIBILITY:
Inclusion Criteria:

* Male / female babies who were born before the mother at the Hacettepe University Children's Hospital Neonatal Intensive Care Unit and / or Hacettepe University Adult Hospital Maternity and Birth Service and were born earlier than 37 weeks.
* Babies who are at the Hacettepe University Children's Hospital Neonatal Intensive Care Unit and / or Hacettepe University Adult Hospital Maternity and Maternity Service, were born earlier than 37 weeks and continue to be followed regularly in the neonatal outpatient clinic.
* Babies whose informed consent was obtained for their participation by the family.

Exclusion Criteria:

* Babies with SGA (birth weight below 10th percentile according to gestational week) by birth weight
* Babies with chromosomal anomalies
* Babies diagnosed with hypoxic ischemic encephalopathy
* Babies who have had major surgical operations (gastrointestinal anomaly, severe necrotizing enterocolitis requiring surgery, major gastrointestinal system anomaly, major congenital heart anomaly, diaphragmatic hernia)
* Babies with exitus in the neonatal period
* Babies who do not continue regular polyclinic follow-up after discharge
* Babies of families who do not comply with the study protocol
* Babies with missing study data

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Group 1: 29 weeks and six days of gestation and earlier Group 2: Those whose gestational age is between 30 weeks and 33 weeks and sixth days Group 3: Those whose gestational age is between 34 weeks and 37 weeks and sixth day
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
the transition time to the most appropriate complementary diet for premature babies | 24 months
  . In the literature, there are not enough studies on the transition time to the most appropriate complementary diet for premature babies. We planned to do this prospective observational study.

SECONDARY OUTCOMES:
Reaching the targeted number of patients | 24 months
  In this time we aim to reach the targeted number of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- See also: complementary feeding — https://pubmed.ncbi.nlm.nih.gov/22555185/
- See also: weaning and complementary feeding in premature babies — https://pubmed.ncbi.nlm.nih.gov/29502384/

DOCUMENTS (1):
  • Study Protocol (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT04499430/Prot_000.pdf